CLINICAL TRIAL: NCT04073745
Title: A Feasibility and Toxicity Analysis of Single Fraction Stereotactic Body Radiation Therapy for Post-Operative Non-Small Cell Lung Cancer
Brief Title: Single Fraction Stereotactic Body Radiation Therapy After Surgery in Treating Patients With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 81919; NCI-2019-04325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 81919 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Positive Surgical Margin; Resected Mass; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Margins of Excision; Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Beginning at least 2 weeks after surgical resection, patients undergo 1 fraction (or 5 fractions every other day if R2 resection of central tumor) of SBRT.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This trial studies the side effects of single fraction stereotactic body radiation therapy after surgery in treating patients with non-small cell lung cancer. Standard radiation for lung cancer involves delivering small doses of daily radiation for several weeks. However, this technique has resulted in inferior outcomes compared to surgery and is associated with damage to surrounding normal lung. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. Giving stereotactic body radiation therapy in fewer treatment sessions (single fraction) may kill tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess feasibility and toxicity of single-fraction stereotactic body radiation therapy (SBRT) in the post-operative setting.

SECONDARY OBJECTIVES:

I. Assess quality of life following post-operative single-fraction SBRT. II. Assess rate of in-field failures.

TERTIARY OBJECTIVES:

I. Assess progression free survival and overall survival following post-operative SBRT for stage III/IV non-small cell lung cancer (NSCLC).

EXPLORATORY OBJECTIVES:

I. Changes in the inflammatory markers.

OUTLINE:

Beginning at least 2 weeks after surgical resection, patients undergo 1 fraction (or 5 fractions every other day if R2 resection of central tumor) of SBRT.

After completion of study treatment, patients are followed up at 5 and 12 weeks and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Has completed curative-intent surgical resection of lung primary with pathologic diagnosis of NSCLC disease, with pathology to include at least 1 of the following:

  * Close (<=2 mm) or Positive surgical margin (R1/R2) or pathologic N2 disease (with or without extracapsular extension [ECE])
* Anatomic pulmonary resection (lobectomy or pneumonectomy) preferred, although sublobar resection is allowed at the discretion of the treating surgeon. Systemic lobe-specific nodal sampling is required. A minimum of 3 N2 stations must be sampled. Selective lymph node dissection should be completed for patients with known N2 disease
* Women of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence)
* Patient or legal representative must be willing and able to participate in protocol requirements, including pre- and post-treatment survey evaluations and clinical assessments
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Contraindication to SBRT

  * This includes the inability to cooperate with any aspect of SBRT such as the inability to lie still and breath reproducibly
* Prior radiation therapy targeting the same area for which radiation treatment is being planned
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which, in the investigator?s opinion, deems the patient unable to participate in enrollment
* Patients who undergo sublobar resection but are unable to undergo appropriate N1 and N2 lymph node sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or greater toxicities | Up to 5 years
  Hospitalization resulting from radiation treatment will be recorded. Any acute (=< 180 days after the end of radiation therapy [RT]) and late (> 180 days after the end of RT) toxicities will be documented using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicity rates will be presented with Clopper-Pearson 90% confidence intervals (alpha = 0.10).
Feasibility of single fraction SBRT | Up to 5 years
  Feasibility will be assessed by the median time to initiation of systemic treatment (TST) following the combination of surgery and stereotactic body radiation therapy (SBRT), as this interval will reflect the probability of completing intended treatment.

SECONDARY OUTCOMES:
Time to initiation of systemic treatment (TST) | From the date of surgery until the date of systemic treatment initiation, assessed up to 5 years
  The proportion of patients who have TST < 8 weeks will be recorded. The median time will be presented with a 90% confidence interval (CI).
Quality of life (QoL) | Up to 5 years
  The QoL scores, from European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and EORTC QLQ Lung Cancer?Specific Module, and cumulative toxicity rates will be compared be at each time-point (starting 5 weeks after SBRT) between tumor locations using the Mann-Whitney U and Fishers exact tests, respectively. Comparisons of QoL scores between time-points will be made using the Wilcoxon signed rank test. All secondary analysis will be conducted at the 10% significance level. The QoL scores will also be examined for time trends and effects of patient characteristics using regression analysis.
In-field failure (IFF) rate | Up to 5 years
  IFF rate will be reported for the total cohort and at 3- and 5-years. The IFF will be monitored using a Bayesian approach. The monitoring will start after 3 patients have received treatment.

OTHER OUTCOMES:
Progression free survival (PFS) | Up to 5 years
  The PFS will be described using standard Kaplan-Meier methodologies. The median survival time, 3-year survival rate, and 5-year survival rate will be estimated and presented with 90% CI.
Overall survival (OS) | From SBRT completion until death (event) or end of study/lost to follow-up (censored), assessed up to 5 years
  The OS will be described using standard Kaplan-Meier methodologies. The median survival time, 3-year survival rate, and 5-year survival rate will be estimated and presented with 90% CI.
Change in immune markers | Baseline up to 5 weeks post-SBRT
  Changes in the mediators of tumor antigen presentation, costimulatory molecules, immune effector cell populations, such as CD4+ and CD8+ T-cells, T regulatory cells (CD4+CD25+FoxP3+), natural killer (NK) cells, monocytes, macrophages, dendritic cells (DCs) and myeloid derived suppressor cells (MDSCs) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States